CLINICAL TRIAL: NCT00424268
Title: Effect of Roflumilast in COPD Patients Treated With Tiotropium. A 24-week, Double-blind Study With 500 µg Roflumilast Once Daily Versus Placebo. The HELIOS Study
Brief Title: Effect of Roflumilast in Chronic Obstructive Pulmonary Disease (COPD) Patients Treated With Tiotropium: The HELIOS Study (BY217/M2-128)
Acronym: HELIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-128; 2006-004508-37 (EudraCT Number)
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): Roflumilast 500 µg
  underlying medication: tiotropium 18 µg, once daily, inhaled
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo
  underlying medication: tiotropium 18 µg, once daily, inhaled
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 µg, once daily, oral administration in the morning
  Arms: Roflumilast
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The aim of the study is to compare the efficacy of roflumilast to placebo on pulmonary function and symptomatic parameters in patients with chronic obstructive pulmonary disease (COPD) during concomitant administration of tiotropium. The study duration will last up to 28 weeks. The study will provide further data on safety and tolerability of roflumilast.

ELIGIBILITY:
Main Inclusion Criteria:

* History of COPD for at least 12 months prior to baseline visit and chronic productive cough for 3 months in each of the 2 years prior to baseline visit
* FEV1/FVC ratio (post-bronchodilator) ≤ 70%
* FEV1 (post-bronchodilator) between ≥ 40% and ≤ 70% of predicted
* Treated with tiotropium for at least 3 months before enrollment
* At least 28 puffs of rescue medication during last week prior to randomization

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticosteroids and/or antibiotics not stopped at least 4 weeks prior to baseline visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (95):
- Austria (5):
  - Altana Pharma/Nycomed Investigational Site, Feldbach
  - Altana Pharma/Nycomed Investigational Site, Gänserndorf
  - Altana Pharma/Nycomed Investigational Site, Hallein
  - Altana Pharma/Nycomed Investigational Site, Linz
  - Altana Pharma/Nycomed Investigational Site, Spittal an der Drau
- France (14):
  - Altana Pharma/Nycomed Investigational Site, Beuvry
  - Altana Pharma/Nycomed Investigational Site, Chauny
  - Altana Pharma/Nycomed Investigational Site, Grasse
  - Altana Pharma/Nycomed Investigational Site, Lyon
  - Altana Pharma/Nycomed Investigational Site, Martigues
  - Altana Pharma/Nycomed Investigational Site, Montigny-lès-Metz
  - Altana Pharma/Nycomed Investigational Site, Nantes
  - Altana Pharma/Nycomed Investigational Site, Nice
  - Altana Pharma/Nycomed Investigational Site, Nîmes
  - Altana Pharma/Nycomed Investigational Site, Ollioules
  - Altana Pharma/Nycomed Investigational Site, Perpignan
  - Altana Pharma/Nycomed Investigational Site, Saint-Laurent-du-Var
  - Altana Pharma/Nycomed Investigational Site, Saint-Quentin
  - Altana Pharma/Nycomed Investigational Site, Toulon
- Germany (16):
  - Altana Pharma/Nycomed Investigational Site, Bad Homburg
  - Altana Pharma/Nycomed Investigational Site, Dortmund
  - Altana Pharma/Nycomed Investigational Site, Geesthacht
  - Altana Pharma/Nycomed Investigational Site, Gelnhausen
  - Altana Pharma/Nycomed Investigational Site, Göppingen
  - Altana Pharma/Nycomed Investigational Site, Hanover
  - Altana Pharma/Nycomed Investigational Site, Koblenz
  - Altana Pharma/Nycomed Investigational Site, Landsberg/Lech
  - Altana Pharma/Nycomed Investigational Site, Leonberg
  - Altana Pharma/Nycomed Investigational Site, Marburg
  - Altana Pharma/Nycomed Investigational Site, Saarbrücken
  - Altana Pharma/Nycomed Investigational Site, Saarlouis
  - Altana Pharma/Nycomed Investigational Site, Schwetzingen
  - Altana Pharma/Nycomed Investigational Site, Sinsheim
  - Altana Pharma/Nycomed Investigational Site, Weyhe
  - Altana Pharma/Nycomed Investigational Site, Witten
- Hungary (10):
  - Altana Pharma/Nycomed Investigational Site, Budapest
  - Altana Pharma/Nycomed Investigational Site, Cegléd
  - Altana Pharma/Nycomed Investigational Site, Csorna
  - Altana Pharma/Nycomed Investigational Site, Érd
  - Altana Pharma/Nycomed Investigational Site, Győr
  - Altana Pharma/Nycomed Investigational Site, Hódmezovásárhely
  - Altana Pharma/Nycomed Investigational Site, Mátraháza
  - Altana Pharma/Nycomed Investigational Site, Nyiregyháza
  - Altana Pharma/Nycomed Investigational Site, Szentes
  - Altana Pharma/Nycomed Investigational Site, Szolnok
- Italy (10):
  - Altana Pharma/Nycomed Investigational Site, Bassano Del Grappa (VI)
  - Altana Pharma/Nycomed Investigational Site, Cisanello (PI)
  - Altana Pharma/Nycomed Investigational Site, Foggia
  - Altana Pharma/Nycomed Investigational Site, Genova
  - Altana Pharma/Nycomed Investigational Site, Milan
  - Altana Pharma/Nycomed Investigational Site, Modena
  - Altana Pharma/Nycomed Investigational Site, Pavullo Nel Frignano (MO)
  - Altana Pharma/Nycomed Investigational Site, Pordenone
  - Altana Pharma/Nycomed Investigational Site, Reggio Emilia
  - Altana Pharma/Nycomed Investigational Site, Verona
- Spain (18):
  - Altana Pharma/Nycomed Investigational Site, A Coruña
  - Altana Pharma/Nycomed Investigational Site, Alicante
  - Altana Pharma/Nycomed Investigational Site, Baracaldo (Vizcaya)
  - Altana Pharma/Nycomed Investigational Site, Candia
  - Altana Pharma/Nycomed Investigational Site, Escaldes-Engordany
  - Altana Pharma/Nycomed Investigational Site, Galdakao
  - Altana Pharma/Nycomed Investigational Site, Guadalajara
  - Altana Pharma/Nycomed Investigational Site, Jerez de la Frontera
  - Altana Pharma/Nycomed Investigational Site, Lleida
  - Altana Pharma/Nycomed Investigational Site, Lugo
  - Altana Pharma/Nycomed Investigational Site, Madrid
  - Altana Pharma/Nycomed Investigational Site, Mostoles Madrid
  - Altana Pharma/Nycomed Investigational Site, Pozuelo de Alarcón
  - Altana Pharma/Nycomed Investigational Site, Requena
  - Altana Pharma/Nycomed Investigational Site, Sant Cugat del Vallès
  - Altana Pharma/Nycomed Investigational Site, Santa Cruz de Tenerife
  - Altana Pharma/Nycomed Investigational Site, Seville
  - Altana Pharma/Nycomed Investigational Site, Valencia
- United Kingdom (22):
  - Altana Pharma/Nycomed Investigational Site, Ashford
  - Altana Pharma/Nycomed Investigational Site, Atherstone, Warwick
  - Altana Pharma/Nycomed Investigational Site, Barry
  - Altana Pharma/Nycomed Investigational Site, Bexhill-on-Sea, East Sussex
  - Altana Pharma/Nycomed Investigational Site, Bolton
  - Altana Pharma/Nycomed Investigational Site, Bolton Lancs
  - Altana Pharma/Nycomed Investigational Site, Chesterfield
  - Altana Pharma/Nycomed Investigational Site, Chesterfield Derbyshire
  - Altana Pharma/Nycomed Investigational Site, Chippenham
  - Altana Pharma/Nycomed Investigational Site, Co. Antrim
  - Altana Pharma/Nycomed Investigational Site, Darlington, Co. Durham
  - Altana Pharma/Nycomed Investigational Site, East Sussex
  - Altana Pharma/Nycomed Investigational Site, Glasgow
  - Altana Pharma/Nycomed Investigational Site, Harrow
  - Altana Pharma/Nycomed Investigational Site, Keresely End, Coventry
  - Altana Pharma/Nycomed Investigational Site, Plymouth
  - Altana Pharma/Nycomed Investigational Site, Sheffield
  - Altana Pharma/Nycomed Investigational Site, Solihull
  - Altana Pharma/Nycomed Investigational Site, Swindon, Wilts
  - Altana Pharma/Nycomed Investigational Site, Trowbridge
  - Altana Pharma/Nycomed Investigational Site, Watford
  - Altana Pharma/Nycomed Investigational Site, Yaxley

REFERENCES:
- [Result] Fabbri LM, Calverley PM, Izquierdo-Alonso JL, Bundschuh DS, Brose M, Martinez FJ, Rabe KF; M2-127 and M2-128 study groups. Roflumilast in moderate-to-severe chronic obstructive pulmonary disease treated with longacting bronchodilators: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):695-703. doi: 10.1016/S0140-6736(09)61252-6. PMID 19716961
- [Derived] Cazzola M, Picciolo S, Matera MG. Roflumilast in chronic obstructive pulmonary disease: evidence from large trials. Expert Opin Pharmacother. 2010 Feb;11(3):441-9. doi: 10.1517/14656560903555201. PMID 20102307

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast: Roflumilast 500 µg, once daily, oral and tiotropium 18 µg, once daily, inhaled
- Placebo: Placebo, once daily, oral and tiotropium 18 µg, once daily, inhaled
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 371 (Includes all randomized patients who took at least one dose of the investigational drug.) | 372 (Includes all randomized patients who took at least one dose of the investigational drug.)
Completed | 309 | 333
Not Completed | 62 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 371 | 372 | 743
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.1) | 64.0 (9.3) | 64.1 (9.2)
Gender [Count of Participants; unit: Participants]
  Female | 109 | 105 | 214
  Male | 262 | 267 | 529

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: Mean change from baseline during the treatment period in pre-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT (Intention to Treat) analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 365 | 364
mL | 65 (12) | -16 (12)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; Repeated measurements analysis (change from baseline over 24 weeks of treatment taking all post-randomization measurements into account); Mean Difference (Net) = 80, 95% CI 2-sided [51 to 110], Standard Error of Mean 15

2. Secondary Outcome: Post-bronchodilator FEV1
Description: Mean change from baseline during the treatment period in post-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 364 | 363
mL | 74 (12) | -7 (11)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 81, 95% CI 2-sided [51 to 110], Standard Error of Mean 15

3. Secondary Outcome: COPD Exacerbation Rate (Moderate or Severe)
Description: Mean rate of COPD exacerbations requiring oral or parenteral glucocorticosteroids (=moderate COPD exacerbations), or requiring hospitalization, or leading to death (=severe COPD exacerbations), per patient per year. A COPD exacerbation is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management [American Thoracic Society (ATS) / European Respiratory Society (ERS) 2005].
Time Frame: 24 weeks treatment period
Population: ITT analysis
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 371 | 372
exacerbations per patient per year | 0.262 [0.184 to 0.375] | 0.342 [0.248 to 0.472]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.1957, Poisson regression — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; Rate ratio = 0.768, 95% CI 2-sided [0.515 to 1.146], Standard Error of Mean 0.157

4. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score
Description: The TDI is a recognized questionnaire to measure dyspnea in an out patient COPD population. At baseline, 3 components of dyspnea, each graded with 4 questions, were asked: - Functional Impairment - Magnitude of Task - Magnitude of Effort At each of the post-randomization visits questions from the TDI were asked related to 3 components: Change in - Functional Impairment - Magnitude of Task - Magnitude of Effort Each question in the TDI is graded from -3 (major deterioration) to +3 (major improvement). This results in a TDI Focal Score ranging from -9 to +9.
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 364 | 364
scores on a scale | 1.4 (0.1) | 0.9 (0.1)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0032, ANCOVA — This secondary endpoint was analyzed in an exploratory manner; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.1 to 0.7], Standard Error of Mean 0.1

5. Secondary Outcome: Shortness of Breath Questionnaire (SOBQ) Total Score
Description: Mean change from baseline during the treatment period in SOBQ. This is a 24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living. The questions were administered at visits V0, V2, V3, V4, V5, V6 and Vend to assess the perceived shortness of breath of the patient. For each activity listed in the questionnaire the patient should rate his/her breathlessness on a scale between zero and five, where zero is "not at all breathless" and five is "maximally breathless or too breathless to do the activity".
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 359 | 359
scores on a scale | -3.4 (0.7) | -0.7 (0.7)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0051, ANCOVA — This secondary endpoint was analyzed in an exploratory manner; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.6, 95% CI 2-sided [-4.5 to -0.8], Standard Error of Mean 0.9

ADVERSE EVENTS:
Time Frame: 24 weeks treatment period
Description: The Safety Set was based on all randomized patients who took at least one dose of the investigational drug after randomization. Three patients randomized to placebo received roflumilast instead and were included in the roflumilast group for safety analyses.
Arm/Group | Roflumilast | Placebo
Serious Adverse Events (participants affected / at risk) | 22/374 | 21/369
Other Adverse Events (participants affected / at risk) | 106/374 | 76/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=374) | Placebo (N=369)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Vascular operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=374) | Placebo (N=369)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 54 (64) | 63 (80) — non-serious
Nasopharyngitis (Infections and infestations) | 21 (24) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 33 (38) | 2 (2)
Weight decreased (Investigations) | 20 (20) | 2 (2) — non-serious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study results may be published and/or presented at scientific meetings. Prior to any submission, all manuscripts/abstracts must be presented to the sponsor for possible comments.